CLINICAL TRIAL: NCT01849146
Title: Phase I Study of AZD1775 (Adavosertib) With Radiation and Temozolomide in Patients With Newly Diagnosed Glioblastoma and Evaluation of Intratumoral Drug Distribution in Patients With Recurrent Glioblastoma
Brief Title: Adavosertib, Radiation Therapy, and Temozolomide in Treating Patients With Newly Diagnosed or Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00858; NCI-2013-00858 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ABTC 1202; ABTC-1202 (Other: Adult Brain Tumor Consortium); ABTC-1202 (Other: CTEP); UM1CA137443 (NIH)
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — adavosertib; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (adavosertib, temozolomide, radiation) (Experimental): INITIATION CYCLE: Patients receive adavosertib PO on days 1, 3, and 5 or 1-5 weekly and temozolomide PO QD for 6 weeks. Patients also undergo concurrent radiation therapy 5 days per week for 6 weeks.
  MAINTENANCE CYCLES: Beginning in week 10, patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Radiation: Radiation Therapy; Drug: Temozolomide
- Arm II (adavosertib, temozolomide) (Experimental): Patients receive adavosertib PO QD on days 1, 3, and 5 or 1-5 weekly, and temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Drug: Temozolomide

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD 1775; AZD-1775; AZD1775; MK 1775; MK-1775; MK1775
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm I (adavosertib, temozolomide, radiation)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I trial studies the side effects and best dose of adavosertib when given together with radiation therapy and temozolomide in treating patients with glioblastoma that is newly diagnosed or has come back. Adavosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving adavosertib, radiation therapy, and temozolomide may work better in treating patients with newly diagnosed or recurrent glioblastoma compared to radiation therapy and temozolomide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated doses (MTD) of AZD1775 (adavosertib) in combination with the current standard of care (radiotherapy/temozolomide for concomitant therapy and temozolomide for adjuvant therapy) for treating patients with newly diagnosed glioblastoma.

II. To define the MTD of AZD1775 (adavosertib) in combination with 6 weeks of daily (Monday-Friday [M-F]) radiotherapy (RT) and concomitant temozolomide (TMZ) administered at 75 mg/m^2/day in patients with newly diagnosed glioblastoma. (Arm 1) III. To define the MTD of AZD1775 (adavosertib) in combination with adjuvant TMZ administered at 150 mg/m^2/day-200 mg/m^2/day for 5 days every 28 days in patients with glioblastoma after concurrent RT/TMZ. (Arm 2)

SECONDARY OBJECTIVES:

I. To characterize the safety profile of AZD1775 (adavosertib) in combination with RT and concomitant TMZ (Arm 1) and AZD1775 (adavosertib) with adjuvant TMZ (Arm 2) in patients with newly diagnosed glioblastoma.

II. To assess the pharmacokinetic (PK) profile of AZD1775 (adavosertib) in combination with upfront radiation/TMZ and adjuvant TMZ in patients with newly diagnosed glioblastoma.

INTRATUMORAL CORRELATIVES/PHARMACOKINETICS OBJECTIVES:

I. To determine the intratumoral concentration of AZD1775 (adavosertib) achieved in patients treated with the putative MTD.

II. To characterize the time course of AZD1775 (adavosertib) in extracellular fluid within brain tumors following a single oral dose of drug by microdialysis.

III. To characterize the pharmacodynamic effects of AZD1775 on tumor through immunohistochemistry (IHC) analysis of pRb (S807/811), proliferation (e.g. Ki-67), pCDC2, Wee1, and apoptosis (e.g. cleaved caspase 3) on resected tumors exposed to drug.

IV. To characterize MGMT methylation and P53 pathway status, also P-gp and wee1 expression levels in patients with newly diagnosed glioblastoma treated with standard therapy in combination with AZD1775 (adavosertib).

V. To explore and analyze adaptive resistance mechanisms to AZD1775 using proteogenomics, and connect this data to spatially resolved drug distribution through targeted, imaging-based quantification of drug efficacy and tumor response.

OUTLINE: This is a dose-escalation study of adavosertib. Patients are assigned to 1 of 2 treatment arms.

ARM I:

INITIATION CYCLE: Patients receive adavosertib orally (PO) on days 1, 3, and 5 or days 1-5 weekly and temozolomide PO once daily (QD) for 6 weeks. Patients also undergo concurrent radiation therapy 5 days per week for 6 weeks.

MAINTENANCE CYCLES: Beginning in week 10, patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive adavosertib PO QD on days 1, 3, and 5 or 1-5 weekly, and temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a tumor tissue form indicating availability of archived tissue from initial resection at diagnosis of glioblastoma completed and signed by a pathologist
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal; if above the institutional upper limit of normal but =< 3 times institutional upper limit of normal, the decision to initiate temozolomide treatment should carefully consider the benefits and risks for the individual patient
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Activated partial thromboplastin time (APTT)/partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
* Patients must be able to provide written informed consent
* Patients must have magnetic resonance imaging (MRI) within 21 days of starting treatment
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry; women of childbearing potential and men must agree to use two birth control methods (either two barrier methods or a barrier method plus a hormonal method) or abstinence prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years
* Patients must be maintained on a stable corticosteroid regimen (no increase for 5 days) prior to the start of treatment
* Patients must be able to swallow whole capsules
* PHASE I PATIENTS:
* Must have histologically proven glioblastoma
* Must have recovered from the immediate post-operative period
* Patients going on Arm 1 or combination dose cohort must not have received prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, tumor infiltrating lymphocytes [TIL], lymphokine-activated killer [LAK] or gene therapy), or hormonal therapy for their brain tumor; glucocorticoid therapy is allowed
* Patients going on Arm 2 must have received planned treatment with radiation therapy and concomitant temozolomide at least 28 days but no more than 49 days prior to starting treatment on this study; patients must have received at least 80% of planned temozolomide and radiation therapy with no grade 3 or grade 4 toxicity (except lymphopenia) attributed to the temozolomide; Arm 2 patients may not have received any other prior chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK or gene therapy), or hormonal therapy for their brain tumor; prior Gliadel wafers are allowed; glucocorticoid therapy is allowed
* INTRATUMORAL DRUG DISTRIBUTION STUDY PATIENTS:
* Patients must have prior histologically proven glioblastoma that is progressive or recurrent following radiation therapy +/- chemotherapy
* Patients must be undergoing repeat surgery that is clinically indicated as determined by their care providers
* Patients must have measurable contrast-enhancing progressive or recurrent glioblastoma by MRI within 21 days of starting treatment; patient must be able to tolerate MRIs
* Patients may have an unlimited number of prior therapy regimens
* Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., Tarceva, hydroxychloroquine, bevacizumab, etc.)

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or AZD1775 (adavosertib) are ineligible; the AZD1775 (adavosertib) investigator brochure and the temozolomide package insert can be referenced for more information
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol; patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs; patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of AZD1775 (adavosertib)
* Patients may not be on drugs known to be moderate or potent inhibitors/inducers of CYP3A4, sensitive substrates of CYP3A4, or substrates of CYP3A4 with narrow therapeutic windows
* Patients may not be on anti-coagulants (warfarin, etc.) other than low-molecular weight heparin (LMWH)
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study because AZD1775 (adavosertib) has potential for teratogenic or abortifacients effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD1775 (adavosertib), breastfeeding should be discontinued if the mother is treated with AZD1775 (adavosertib)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD1775 (adavosertib); in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of adavosertib with 6 weeks of radiotherapy and temozolomide (Arm I) | Up to 6 weeks
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Severity and frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportion of subjects who experience grade 3 or above toxicities will be estimated, along with 95% confidence intervals by each type of toxicity.
Maximum tolerated dose of adavosertib with adjuvant temozolomide (Arm II) | Up to 28 days
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Severity and frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportion of subjects who experience grade 3 or above toxicities will be estimated, along with 95% confidence intervals by each type of toxicity.
Incidence of toxicities | Up to 30 days post-treatment
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Severity and frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportion of subjects who experience grade 3 or above toxicities will be estimated, along with 95% confidence intervals by each type of toxicity.

SECONDARY OUTCOMES:
Overall survival | The time from the date of initial diagnosis to the date of death, assessed up to 2 years
  Calculated using the Kaplan-Meier method.
Progression-free survival | The time from the date of initial diagnosis to the date progressive disease was defined and also patient was alive, assessed up to 2 years
  Calculated using the Kaplan-Meier method.

OTHER OUTCOMES:
Pharmacokinetic profile of adavosertib in combination with radiation and temozolomide and adjuvant temozolomide | Baseline, at 0.5, 1, 2, 4, 6, 8 and 24 hours of weeks 1 and 4 of cycle 1 (Arm I) and at baseline, 0.5, 1, 2, 4, 6, 8, and 24 hours of cycle 1 (Arm II)
  Individual subject plasma concentration-time curves will be analyzed by non-compartmental methods using routines supplied in the WinNonlin Professional Version 5.0 software package (Pharsight Corp., Cary, North Carolina). The geometric mean +/- standard deviation of the estimated values of the pharmacokinetic parameter for groups of subjects evaluated at maximum tolerated dose level will be calculated. Parametric statistical tests (i.e., single factor analysis of variance, Student's t-test) of pharmacokinetic variables will be performed after logarithmic transformation of the data.
Intratumoral adavosertib concentration | Up to the day of surgery
  Will be summarized using descriptive statistics.
pRb (S807/811) expression levels | Up to 2 years
  Will be summarized using descriptive statistics.
Proliferation (Ki-67) expression levels | Up to 2 years
  Will be summarized using descriptive statistics.
pCDC2 expression levels | Up to 2 years
  Will be summarized using descriptive statistics.
Apoptosis (cleaved caspase 3) levels | Up to 2 years
  Will be summarized using descriptive statistics.
Genotyping data | Up to 2 years
  Will be summarized using descriptive statistics.
MGMT methylation status | Up to 2 years
  Will be summarized using descriptive statistics.
P53 mutation status | Up to 2 years
  Will be summarized using descriptive statistics.
P-gp expression level | Up to 2 years
  Will be summarized using descriptive statistics.
Wee1 expression level | Up to 2 years
  Will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Eudocia Q Lee, Principal Investigator — National Cancer Institute (NCI)
Locations (12):
- United States (12):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania